CLINICAL TRIAL: NCT04381052
Title: A Randomized Placebo-Controlled Safety and Dose-Finding Study for the Use of the IL-6 Inhibitor Clazakizumab in Patients With Life-threatening COVID-19 Infection
Brief Title: Study for the Use of the IL-6 Inhibitor Clazakizumab in Patients With Life-threatening COVID-19 Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to poor enrollment. Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1).
Sponsor: Columbia University (Other)
Collaborators: NYU Langone Health (Other); CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAT0142
Record Dates: First submitted 2020-05-06; First posted 2020-05-08 (Actual); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: Coronavirus; SARS-COVID-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — clazakizumab

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, adaptive seamless Phase II/III design (ASD). The investigators propose the administration of an investigational drug in patients with high predicted short-term mortality secondary to COVID-19 disease. Patients will be enrolled and randomly assigned in a 1:1 ratio to two study arms that will receive clazakizumab at a dose of 25 mg or placebo.
Who Masked: Participant, Investigator
Masking Description: This study is double-blind and therefore neither the Investigator, the subject, the Sponsor and its representatives, nor other designated study site personnel involved in running of the study will be aware of the identification of the investigational drug administered to each subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clazakizumab 25 mg (Experimental): The first dose will be administered as soon as possible after the patient is enrolled and randomized into the Clazakizumab 25 mg arm. The route of administration will be intravenous. Each dose will be administered as an infusion that is run over 30 minutes. Serum C-reactive protein (CRP) will be evaluated at baseline and on days 1 and 2 following clazakizumab administration. If the CRP does not decrease by 50% within 36-48 hours after the first dose, a second dose of 25 mg clazakizumab will be given no later than day 3.
  Interventions: Drug: Clazakizumab
- Placebo (Placebo Comparator): The first dose will be administered as soon as possible after the patient is enrolled and randomized into the Placebo arm. The route of administration will be intravenous. Each dose will be administered as an infusion that is run over 30 minutes. Serum CRP will be evaluated at baseline and on days 1 and 2 following clazakizumab administration. If the CRP does not decrease by 50% within 36-48 hours after the first dose, a second dose of placebo will be given no later than day 3.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Clazakizumab — Dose is 25mg intravenously over 30 minutes.
  Other Names: Clazakizumab solution
  Arms: Clazakizumab 25 mg
Other: Placebo — Intravenously administered over 30 minutes.
  Arms: Placebo

SUMMARY:
In this study, the investigators propose to administer clazakizumab to patients with life-threatening Coronavirus Disease 2019 (COVID-19) infection manifest by pulmonary failure and a clinical picture consistent with a cytokine storm syndrome. This is a single-center randomized, double-blind, placebo-controlled trial in which 30 patients will be enrolled and randomly assigned in a 1:1 ratio to two study arms and receive clazakizumab at a dose of 25 mg or placebo.

DETAILED DESCRIPTION:
The limited understanding of the clinical behavior of patients infected with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) (the viral organism responsible for COVID-19 disease) is evolving on a daily basis. Reports from China indicate that a subset of patients with the worst clinical outcomes may manifest cytokine storm syndrome. Hypotheses that excess cytokines may trigger a secondary hemophagocytic lymphohistiocytosis (sHLH) have been proposed. Indeed, cytokine profiles consistent with this picture were observed in Chinese patients with severe pulmonary involvement. Specifically, elevated ferritin and interleukin-6 (IL-6) were associated with fatalities among the infected patients. A role for targeted anti-inflammatory and anti-cytokine therapies in the treatment of pulmonary hyperinflammation has been proposed.

Clazakizumab is a genetically engineered humanized immunoglobulin-1 (IgG1) monoclonal antibody (mAb) that binds with high affinity to human IL-6. This investigational agent is currently being studied as a treatment for chronic active antibody mediated rejection of renal allografts.

In this study investigators propose to administer clazakizumab to patients with life-threatening pulmonary failure secondary to COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, the patients must meet all of the following criteria:

1. At least 18 years of age
2. Confirmed COVID-19 disease (by Cobas SARS-CoV-2 real time reverse transcription polymerase chain reaction (RT-PCR) using nasopharyngeal swab sample, or equivalent test available to be performed by the Columbia University Irving Medical Center (CUIMC)/New York Presbyterian (NYP) clinical laboratory). Effort will be made to have the confirmatory test result <72 hours prior to enrollment however given overall clinical demand this may not be feasible in all cases.
3. Respiratory failure manifesting as: Acute Respiratory Distress Syndrome (defined by a P/F ratio of <200), OR oxygen saturation (SpO2) < 90% on 4 liters (L) (actual or expected given higher O2 requirement) OR increasing O2 requirements over 24 hours, plus 2 or more of the following predictors for severe disease:

   CRP > 35 mg/L Ferritin > 500 ng/mL D-dimer > 1 mcg/L Neutrophil-Lymphocyte Ratio > 4 Lactate dehydrogenase (LDH) > 200 U/L Increase in troponin in patient w/out known cardiac disease
4. Has a consent designee willing to provide informed consent on behalf of the patient (this assumes that a mechanically ventilated patients lacks capacity to consent on his/her own behalf. Should it be deemed that the patient has capacity to consent, consent may be obtained from the patient.)
5. Women of childbearing potential must be willing and able to use at least one highly effective contraceptive method for a period of 5 months following the study drug administration. In the context of this study, an effective method is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly such as:

   1. combined (estrogen and progestogen containing) hormonal contraception combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, or transdermal)
   2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
   3. intrauterine device (IUD)
   4. intrauterine hormone-releasing system (IUS)
   5. vasectomized partner
   6. bilateral tubal occlusion
   7. true abstinence. when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence, such as calendar, ovulation, symptothermal, postovulation methods, and withdrawal are not acceptable methods of contraception.
6. Men must be willing to use a double-barrier contraception from enrollment until at 5 months after the last dose of study drug, if not abstinent.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Evidence of irreversible injury deemed non-survivable even if the pulmonary failure recovers (for example severe anoxic brain injury)
2. Known active inflammatory bowel disease
3. Known active, untreated diverticulitis
4. Known untreated bacteremia
5. Pregnancy. (The protocol will exclude pregnant subjects given the lack of overall data on use of clazakizumab in pregnancy however the study team would consider a protocol revision should more than 3 potential pregnant study subjects be excluded on this basis).
6. Known hypersensitivity to the clazakizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Cohen, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center / New York Presbyerian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Coded data will be shared with New York University (NYU) Langone for the purpose of statistical analysis and scientific reporting.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was closed due to no further development. Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1). Assignment was not unblinded/disclosed.
Groups:
- Clazakizumab 25 mg or Placebo: The first dose will be administered as soon as possible after the patient is enrolled and randomized into a specific arm. The route of administration will be intravenous. Each dose will be administered as an infusion that is run over 30 minutes. Serum CRP will be evaluated at baseline and on days 1 and 2 following first dose administration. If the CRP does not decrease by 50% within 36-48 hours after the first dose, a second dose of placebo will be given no later than day 3.
  Placebo: Intravenously administered over 30 minutes. OR Clazakizumab: Dose is 25mg intravenously over 30 minutes.
Period: Overall Study
Arm/Group | Clazakizumab 25 mg or Placebo
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Study was closed due to no further development. Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1). Assignment was not unblinded/disclosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clazakizumab 25 mg | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Serious Adverse Events Associated With Clazakizumab or Placebo
Time Frame: 60 days
Population: Study stopped due to no further development. Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1). Assignment was not unblinded/disclosed.
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Cumulative Incidence of Intubation
Time Frame: 14 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Extubation
Time Frame: 14 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Length of Intensive Care Unit (ICU) Stay
Time Frame: 14 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Patients Who Present a Decrease in C-reactive Protein (CRP)
Time Frame: 14 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Patients With Acute Kidney Injury (AKI)
Time Frame: 14 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Patients With a Need for Renal Replacement Therapy (RRT)
Time Frame: 14 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Duration of Renal Replacement Therapy (RRT)
Time Frame: 60 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Patient Survival
Description: Number of participants alive at day 28.
Time Frame: 28 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Patient Survival
Description: Number of participants alive at day 60, end of study.
Time Frame: 60 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Patients With Hemodialysis
Time Frame: 60 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Patients With Continuous Renal Replacement Therapies (CRRT)
Time Frame: 60 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Patients With Peritoneal Dialysis
Time Frame: 60 days
Population: as for outcome 1
Arm/Group | Clazakizumab 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 60 days
Description: Study stopped due to no further development. Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1). Assignment was not unblinded/disclosed.
Arm/Group | Clazakizumab 25 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study was closed due to no further development. Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1). Assignment was not unblinded/disclosed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT04381052/Prot_SAP_000.pdf